CLINICAL TRIAL: NCT06974318
Title: The Evaluation of the Effect of ABCDEF Bundle Implementation on Preventing Delirium in Patients Followed in the Medical Intensive Care Patients Due to Chronic Obstructive Pulmonary Disease
Brief Title: ABCDEF Bundle to Prevent Delirium for COPD Patients
Acronym: COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Emine Ezgi Ozcelik, Nurse, MSc, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IstanbulSBU-HSBE-EEO-01
Record Dates: First submitted 2025-04-22; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Delirium; Copd; Nurse's Role
MeSH Terms: conditions — Delirium; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: A-Two Arms Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Other): This group will have "Standart Nursing Care" to prevent delirium.
  Interventions: Other: Standard Care to Prevent Delirium
- Intervention Group (Experimental): This group will have "ABCDEF Bundle" to prevent delirium.
  Interventions: Other: ABCDEF Bundle to Prevent Delirium

INTERVENTIONS:
Other: ABCDEF Bundle to Prevent Delirium — The ABCDEF Care Bundle-comprising components focused on pain management (A), spontaneous awakening and breathing trials (B), choice of sedation and analgesia (C), delirium assessment and management (D), early mobility (E), and family engagement (F)-was developed to promote patient-centered care in the ICU and improve clinical outcomes. Nurses play a central role in the effective implementation of this bundle, given their continuous patient interaction and responsibility for early detection and response to delirium symptoms.
  Arms: Intervention Group
Other: Standard Care to Prevent Delirium — Standard care inclued pain management, Glasgow Coma Scale evaluation, Richmond Agitation-Sedation Scale evaluation and control of the stimulations.
  Arms: Control Group

SUMMARY:
Abstract Chronic Obstructive Pulmonary Disease (COPD) is a progressive respiratory disorder characterized by persistent airflow limitation and chronic respiratory symptoms, resulting from abnormalities in the bronchi, bronchioles, and alveoli. Patients with COPD may require admission to intensive care units (ICUs), particularly during acute exacerbations. In this context, both disease management and the prevention of potential complications, such as delirium, are of critical importance. Delirium is a common, preventable, and serious complication in ICUs that prolongs hospital stays, increases healthcare costs, and heightens the risk of infections. Hypoxia-induced cognitive impairment is among the key contributing factors to delirium in patients with COPD.

To improve patient outcomes, the ABCDEF Care Bundle was introduced in 2013 as a structured and evidence-based approach to ICU care. This study aims to evaluate the effectiveness of the ABCDEF Care Bundle in preventing delirium in patients with COPD admitted to the ICU. The research will be conducted as a randomized controlled trial between April and December 2025 in the third-level ICU of Taksim Training and Research Hospital. The study population will consist of COPD patients, with a total sample size of 84 patients (42 in each group), randomly assigned using a computer-assisted simple randomization method. A variety of validated instruments will be used to assess pain, sedation, cognitive status, mobility, and sleep quality.

The findings of this study are expected to contribute to the growing body of evidence supporting structured ICU care and to raise awareness among healthcare professionals regarding the implementation of the ABCDEF Care Bundle.

Keywords:

ABCDEF Care Bundle, Delirium, COPD, Intensive Care, Nursing Care, Randomized Controlled Trial

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over,
* No cognitive disease such as dementia or Alzheimer's,
* Patients requiring intensive care monitoring for at least 24 hours,
* Non-intubated patients,
* Having a diagnosis of COPD.

Exclusion Criteria:

* Patients being monitored in intensive care primarily due to central nervous system disease,
* Intubated patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The research has not started yet. Instutional (hospital) permission is being awaited. | 12 months
  After obtaining the necessary permissions, data will be collected with forms. Data will be analyzed in the SPSS 29.0 program. Thirteen forms will be used to collect data:
  * Informed Consent Form
  * Patient Information Form
  * Numeric Pain Rating Scale
  * Facial Pain Rating Scale
  * Glasgow Coma Scale
  * Richmond Agitation-Sedation Scale
  * Chronic Obstructive Pulmonary Diseases (COPD) Assessment Questionnaire
  * Nursing Delirium Screening Scale
  * Intensive Care Delirium Control Screening List
  * Richards-Campbell Sleep Questionnaire
  * Intensive Care Unit Mobilization Scale ABCDEF Bundle Action Plan Form ABCDEF Bundle Checklist
  Note: ABCDEF Bundle is included in the literature with this name. This is not an abbreviation. ABCDEF Bundle:
  A: Assess the pain B: Both control spontaneous breathing and awakeaning C: Choice of sedation D: Delirium assesment E: Early mobilization F: Family encouragement and empowerment
  ABCDEF Bundle is working with "all or nothing" rule, so there is no minimum-maximum value.
Power Analysis | 12 months
  The aim of this study was to determine the effectiveness of the ABCDEF care bundle in preventing the development of delirium in COPD patients.The universe of the study will consist of patients who are being followed up with a diagnosis of COPD in the Intensive Care Unit of a Training and Research Hospital. There will be two groups in the study and the differences between the groups will be examined. In line with this study, when the effect level is determined as 0.8 and the power of the test is determined as 0.95, the number of samples that should be reached with a 5% error rate is calculated with the G*Power 3.1.9.4 program, and it has been concluded that a minimum of 42 patients for each group and a total of 84 patients will be included in the study.
Forms- Informed Consent Form | 12 months
  -Informed Consent Form
  The research will be explained verbally to the volunteers participating in the study and both verbal and written consent will be obtained.
Forms- Patient Information Form (1) | 12 months
  -Patient Information Form
  Patients demographic essentials: Gender, age, weight, height (weight and height will be combined to report BMI kg/m²) Marital status: Single, married, divorced, in relationship, unmarried. Education situation: Gratuation of elementery school, high school, collage. Work situation: worker, white collar, retired, unemployee.
  Economic situation: income less than/equal to/more than expenses,
  These questions aim to detect patients worries (economic, work, family), and make nurses alert to their delirium predispositions.
Forms- Patient Information Form (2) | 12 months
  Diagnose date of COPD: How many years with this illness? GOLD degree of COPD: Degree of COPD seriousness. Degree 0-4 and worse when the degree rise.
  APACHE II Score: Predict of critical care mortality. Other diseases: Diabetes mellitus, hypertension. Use of sedation: Benzodiazepines, hypnotics Laboratory results: Arterial blood gas (PaCO2, PaO2, pH, SpO2, base excess), creatinine, CRP, potassium)
  These questions aim to detect prognosis of patient.
  Vital signs: Blood pressure (mmHg), heart rate (minute), respiratory rate (minute), SpO2 (%), temperature (C) Medications: Inotropic medications, antiboitics, inhalers, fluid support, electrolytes, mucolitics, analgesics, antiemetics
  These questions aim to get informed about treatment and make nurses alert about complications (e.g. some antiemetics trigger delirium, hyperthermia can cause change of conscious)
Forms- Chronic Obstructive Pulmonary Disease (COPD) Assessment Questionnaire | 12 months
  -Chronic Obstructive Pulmonary Disease (COPD) Assessment Questionnaire (To assess degree of COPD seriousness) (Necessary permissions have been obtained) The COPD Assessment Test (CAT) is a validated, patient-completed questionnaire designed to evaluate the impact of chronic obstructive pulmonary disease (COPD) on a patient's health status. It consists of 8 items, each scored from 0 to 5, addressing symptoms such as cough, sputum production, chest tightness, breathlessness, and the effect of COPD on daily activities and energy levels. The total score ranges from 0 to 40, with higher scores indicating greater disease impact. The CAT is widely used in clinical practice to support disease management and monitor treatment effectiveness.
Forms- Numeric Pain Rating Scale and Facial Pain Rating Scale | 12 months
  * Numeric Pain Rating Scale (To assess pain whom can communicate) Evaluation is conducted in patients who are able to communicate, and the patient provides a response. A score ranging from 1 to 10 is assigned, where a score of 1 indicates no pain, and a score of 10 represents the highest level of pain.
  * Facial Pain Rating Scale (To assess pain whom can not communicate) Evaluation is conducted based on the facial expression of patients who are unable to communicate. A pain scale from 0 to 5 is used, where a score of 0 indicates no pain, and a score of 5 represents a wrinkled, sweaty facial expression indicative of the highest level of pain.
  It is used as part of the assessment for option "A: Assess the pain" in the ABCDEF bundle.
Forms- Glasgow Coma Scale | 12 months
  -Glasgow Coma Scale (To assess consciousness and awarenes) The Glasgow Coma Scale is a clinical tool used to assess a patient's level of consciousness, particularly following head injuries or neurological impairments. It evaluates three parameters: eye opening, verbal response, and motor response, each scored on a scale.
  The total score ranges from 3 (indicating deep coma or death) to 15 (indicating full consciousness). The tool helps clinicians objectively determine the severity of neurological impairment and monitor patient progress."
  he purpose of using this scale is to provide information about the patient's level of consciousness. It is used as part of the assessment for option "B: Both spontaneous awakening and spontaneous breathing trials" in the ABCDEF bundle.
  Note: Since intubated patients will not be included in the study, an additional form for evaluating spontaneous breathing will not be used.
Forms- Richmond Agitation-Sedation Scale | 12 months
  -Richmond Agitation Sedation Scale (Status of being sedatized) (Necessary permissions have been obtained) The Richmond Agitation-Sedation Scale (RASS) is a clinical tool used to assess a patient's level of sedation or agitation, commonly in critical care settings. It includes 10 levels, ranging from -5 (deep sedation) to +4 (combative agitation). Scores from -5 to -1 indicate varying degrees of sedation, while scores from +1 to +4 represent increasing levels of agitation. The RASS helps healthcare providers guide sedation management and monitor patient comfort and safety.
  The purpose of using this scale is to ensure that nurses remain alert to the patient's level of agitation and sedation. It is employed as part of the assessment for option "C: choice analgesia and sedation" in the ABCDEF bundle.
Forms- Nursing Delirium Screening Tool | 12 months
  -Nursing Delirium Screening Tool (Delirium assessment scale) (Necessary permissions have been obtained) The Nursing Delirium Screening Tool (Nu-DESC) is a brief, nurse-administered instrument designed to detect early signs of delirium in hospitalized patients. It consists of five items-disorientation, inappropriate behavior, inappropriate communication, illusions/hallucinations, and psychomotor retardation-each scored from 0 to 2. A total score of 2 or more suggests the presence of delirium. The Nu-DESC is widely used in clinical settings due to its ease of use, reliability, and effectiveness in facilitating early intervention. It is used as part of the assessment for option "D: Delirium Assessment" in the ABCDEF bundle.
Forms- Intensive Care Delirium Screening List | 12 months
  -Intensive Care Delirium Screening List (Delirium assessment scale) (Necessary permissions have been obtained) The Intensive Care Delirium Screening Checklist (ICDSC) is a validated tool developed to systematically assess delirium in critically ill patients within intensive care units. The checklist comprises 8 items reflecting key diagnostic features of delirium, including altered consciousness, inattention, disorientation, hallucinations, and sleep-wake cycle disturbances. Each item is scored as 0 (absent) or 1 (present), with a total score ranging from 0 to 8. A score of 4 or more indicates the presence of delirium. The ICDSC is widely utilized for regular monitoring, supporting early detection and timely management of delirium in ICU settings. It is used as part of the assessment for option "D: Delirium Assessment" in the ABCDEF bundle.
Forms- Richards-Campbell Sleep Questionnaire | 12 months
  -Richards-Campbell Sleep Questionnaire (Sleep quality assessment scale) (Necessary permissions have been obtained) The Richards-Campbell Sleep Questionnaire (RCSQ) is a validated, patient-reported instrument designed to assess perceived sleep quality in critically ill patients, particularly those in intensive care units. It consists of five visual analog scale items that evaluate sleep depth, latency, number of awakenings, return to sleep, and overall sleep quality. Each item is scored from 0 to 100 mm, with higher scores indicating better sleep. The RCSQ is widely used in clinical research and practice to evaluate sleep disturbances and guide interventions in ICU settings. It is used as part of the assessment for option "D: Delirium Assessment" in the ABCDEF bundle because sleep patterns and disturbances play a significant role in the development of delirium.
Forms- Intensive Care Unit Mobilization Scale | 12 months
  -Intensive Care Unit Mobilization Scale (Level of mebilization scale in ICU) (Necessary permissions have been obtained) The Intensive Care Unit Mobilization Scale (IMS) is a structured tool used to evaluate the level of physical mobilization in critically ill patients within the ICU. It categorizes mobilization into 8 levels, ranging from 0 (no mobilization) to 7 (walking independently). The scale allows clinicians to document and monitor patient progress, facilitate early mobilization efforts, and promote functional recovery. The IMS is widely used in both clinical practice and research to standardize mobilization assessment and support rehabilitation strategies in intensive care settings. It is used as part of the assessment for option "E: Early Mobilization" in the ABCDEF bundle.
Forms- ABCDEF Bundle Action Plan Form | 12 months
  ABCDEF Bundle Action Plan Form This is an action plan form when pain occurs, consciousness/awareness changes, sedation status changes, delirium score rising, mobilization status, family engagement status. As a nurse what can I do?
Forms: ABCDEF Bundle Action Plan Form Explanation (1) | 12 months
  ABCDEF Bundle Action Plan Form
  A: Assess the pain: Pain will be assessed with the appropriate scale at most every four hours. If medication has been administered to a patient with pain, pain will be assessed again after 15-30 minutes and then hourly, depending on the duration of effect of the medication. If it is a noninvasive procedure, pain will be assessed after 30 minutes and hourly.
  B: Both spontaneous breathing and awakening: Invasive ventilated patients will not be allowed to this research, so spontaneous breathing will not be assessed with any scale. Awakeaning will be assessed with Glasgoe Coma Scale.
  C: Choice of sedations: The patient's sedation status will be checked. If the patient is receiving sedation, the type (benzodiazepine etc.) will be recorded. The time when ongoing sedations are stopped will also be recorded. Sedation status will be assessed with the Richmond Agitation-Sedation Scale.
Forms: ABCDEF Bundle Action Plan Form Explanation (2) | 12 months
  ABCDEF Bundle Action Plan Form
  D: Delirium assessment: Delirium will be checked with two scales: Nursing Delirium Screening Tool (Three times a day) and Intensive Care Delirium control Screening Checklist (Two times a day).
  E: Early mobilization: Early mobilization is important for COPD patients. If it is not contraindicated patients will be mobilized at least once a day. Status of mobilization will be determined with Early Mobilization Scale.
  F: Family engagement: Family visits and participation in care are important to prevent delirium from developing in intensive care patients. Since there is no form for this in the literature, the patient will be provided with interaction with the patient's relative at least once a day for at least 15 minutes.
Forms- ABCDEF Bundle Checklist | 12 months
  ABCDEF Bundle Checklist
  This form is an only checklist, no any actions. For example:
  A: Assess the pain: (Check) B: Both spontaneous breathing and awakening: (Check) C: Choice of sedations: (Check) D: Delirium assessment (Check) E: Early mobilization (Check) F: Family engagement (Check)
  Note: The elements within a care bundle represent evidence-based best practices. In routine clinical practice, these elements may not always be implemented consistently, which can lead to variability in patient care. A care bundle aims to combine these practices into a standardized set that should be applied uniformly to every patient, every time.